CLINICAL TRIAL: NCT05151211
Title: Investigation of the Use of 1 Minute Sit to Stand Test to Evaluate Physical Capacity and Effort-Related Desaturation in Individuals With Amyotrophic Lateral Sclerosis
Brief Title: Use of 1 Minute Sit to Stand Test for Physical Capacity and Effort Related Desaturation in Amyotrophic Lateral Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Asena Yekdaneh, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: Gulnergiz
Record Dates: First submitted 2021-11-13; First posted 2021-12-09 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Physical capacity; Desaturation; Dyspne
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validity and Reliability Group: In order to evaluate the usability of the 1 MSTS, the validity and reliability of the test will be examined. In order to determine its validity in assessing physical capacity, the correlation of 1 minute sit up and 6 MWT and quadriceps muscle strength; In order to determine its validity in the evaluation of effort-induced desaturation, the correlation between the change in oxygen saturation and heart rate parameters before and after the 6 MWT and the change before and after the 1 MSTS test will be examined. In order to determine the reliability of the 1 MSTS, a re-test will be performed and 1 MSTS will be applied again after 1 week and the intraclass correlation coefficient will be checked.

SUMMARY:
The aim of this study is to investigate the usability of the 1 Minute Sit to Stand Test (1 MSTS) in evaluating physical capacity and effort-related desaturation in individuals with Amyotrophic Lateral Sclerosis (ALS). In this context, patients diagnosed with ALS who meet the inclusion criteria will be included in the study. For the physical capacity assessment of patients with ALS at different ambulatory levels included in this study, a 6 minutes walking test (6 MWT) and a 1 MSTS will be applied. Before and at the end of the test, the severity of dyspnea and leg fatigue of the patients will be determined by the Modified Borg Scale; effort-induced desaturation and heart rate by fingertip pulse oximetry; peripheral muscle strength (for the quadriceps femoris muscle) will be evaluated with a hand held dynamometer. When the studies are examined, it has been determined that the 6 MWT is relatively difficult to tolerate in individuals with ALS, it may be difficult to provide the necessary space and equipment for the test, and a shorter, easy-to-apply, and practical evaluation method that can be used instead of this test in the clinic is needed. As a result of this study, the usability of the 1 MSTS in individuals with ambulatory ALS in evaluating physical capacity and desaturation due to effort will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS
* 18 years and over
* Ambulatory
* Volunteer to participate in the study

Exclusion Criteria:

* Having a comorbidity that may affect the results of the study (orthopedic, cardiopulmonary, orthopedic, psychiatric, etc.)
* Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with ALS who come to Bakırköy Psychiatric Hospital, Neurology Clinic and meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale (ALSFRS) | Time Frame: Baseline
  ALSFRS, which is used to evaluate the functional status of individuals with ALS, is a scale consisting of 12 parameters: speech, salivation, swallowing, handwriting, feeding, dressing and self-care, turning and covering in bed, walking, climbing stairs, dyspnea, orthopnea and respiratory failure. And evaluated out of a total of 48 points. Each question is scored between 0 and 4 points. While the functionally normal patient gets four points, the scores decrease from four depending on the functional deterioration and zero point is given to the worst functional condition. In this study, the functional levels of the participants will be evaluated with this scale.
1 Minute Sit to Stand Test (1MSTS) | Time Frame: Baseline
  1MSTS will be administered using an armless chair (height = 43 cm). Participants will be asked to sit and stand as quickly and safely as possible for one minute from the time the time starts. The number of times to get out of the chair completed in one minute will be counted and recorded as the test result. In this study, the functionality of the participants will be evaluated with this test.
6 Minutes Walking Test (6MWT) | Time Frame: Baseline
  The 6MWT is a submaximal exercise test used to evaluate aerobic capacity and endurance. The distance traveled during the test is used as an outcome measure to determine physical capacity. In this context, an area of 30 meters long will be determined with cones, and the participants will be asked to walk the maximum distance they can walk between two cones for six minutes. At the end of each minute, a standardized notification will be given, reminding the remaining time and instructing to continue. After six minutes, the total distance walked will be recorded in meters. The greater the distance walked, the greater the test result. In this study, the physical capacity of the participants will be evaluated with this test.
Modified Borg Scale (MBS) | Time Frame: Baseline
  It will be used to evaluate dyspnea and lower extremity muscle fatigue of individuals with ALS before and after the 6 minute walking test and 1 minute sit to stand test. MBS is a scale that is frequently used to evaluate the severity of dyspnea on exertion and severity of dyspnea at rest. It consists of ten items describing the severity of dyspnea according to their degrees.It is similarly used to determine lower extremity fatigue; zero indicates no fatigue in the lower extremities, while the person experiencing maximal fatigue gets 10 points.
Heart Rate Measurement | Time Frame: Baseline
  Before and after the 6 minute walking test and 1 minute sit to stand test, heart rate of the participants will be evaluated with by pulse oximetry. A pulse oximeter is a small, lightweight device used to monitor the amount of oxygen carried in the body and also heart rate. Heart rate, is the number of times the heart beats per minute. A normal resting heart rate should be between 60 to 100 beats per minute. Lower than 60 and higher than 100 can indicate heart rate anomaly.
Quadriceps Muscle Strength | Time Frame: Baseline
  Quadriceps muscle strength will be evaluated bilaterally using a hand held dynamometer. Measurements were to be repeated 2 times in the manual muscle test position and with adequate rest intervals, with the highest value recorded in pounds (lbs). In this study, the quadriceps muscle strength of the participants will be evaluated with this test.
Dyspnea ALS 15 (DALS-15) | Time Frame: Baseline
  The DALS-15 is a one-dimensional scale developed to assess shortness of breath in ALS patients. It can be applied very quickly and easily. The questionnaire consists of 15 questions that the patient can easily answer on their own. The patient expresses his/her condition in the last 2 weeks using a 3-point Likert scale (0=never, 1=occasionally, and 2=often). The total score ranges from 0 (no dyspnea) to a maximum of 30 (severe dyspnea). The higher the score, the greater the severity of dyspnea. In this study, the shortness of breath status of the participants will be evaluated with this scale.
Oxygen Saturation Measurement (SpO2 Measurement) | Time Frame: Baseline
  Before and after the 6 minute walking test and 1 minute sit to stand test, the SpO2 of the participants will be evaluated with by pulse oximetry. A pulse oximeter is a small, light weight device used to monitor the amount of oxygen carried in the body and also heart rate. This non invasive tool will be attached painlessly to paticipants fingertip, sending two wave lengths of light through the finger to measure paticipants heart rate and how much oxygen is in the system. An oxygen saturation level of 95 percent is considered typical for most healthy people. Lower than this percent can indicate low level of oxygen in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Gökşen KURAN ASLAN, Asst. Prof., Study Director — Istanbul University - Cerrahpasa; İrem Kurt, Pt., MSc., Principal Investigator — Istanbul University - Cerrahpasa; Tuğba Akgüller, Pt., MSc., Principal Investigator — Istanbul University - Cerrahpasa; Feray Güngör, Pt., MSc., Principal Investigator — Istanbul University - Cerrahpasa; Nazlı Güngör, Pt., MSc., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No